CLINICAL TRIAL: NCT00803270
Title: Mixed Incontinence: Medical Or Surgical Approach?
Acronym: MIMOSA
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Feasibility Period ended.
Sponsor: Carelon Research (Other)
Collaborators: University of Alabama at Birmingham (Other); University of California, San Diego (Other); University of Maryland (Other); University of Pittsburgh (Other); University of Texas (Other); The University of Texas at San Antonio (Other); University of Utah (Other); Beaumont Hospital (Other); Loyola University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MIMOSA (terminated)
Record Dates: First submitted 2008-12-04; First posted 2008-12-05 (Estimated); Results first posted 2012-05-11 (Estimated); Last update posted 2013-05-10 (Estimated); Status verified 2013-05

CONDITIONS: Urinary Incontinence
Keywords: Stress urinary incontinence, Mixed, Urge
MeSH Terms: conditions — Urinary Incontinence; Urinary Incontinence, Stress | interventions — Surgical Procedures, Operative

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Surgical Treatment (Active Comparator): Surgical treatment will consist of the following evidence-based stress incontinence procedures: mid-urethral slings (TVT, TOT, TVT-O), fascial slings, and Burch colposuspension.
  Interventions: Procedure: Surgical
- Non Surgical Treatment (Active Comparator): The non-surgical treatment will include two components:
  1. Pharmacological therapy with any FDA approved overactive bladder (OAB) drug in approved doses; and
  2. Behavioral therapy.
  Interventions: Drug: Non-Surgical Intervention

INTERVENTIONS:
Drug: Non-Surgical Intervention — Both oral urge incontinence medication and behavioral treatment
  Other Names: Non-Surgical Treatment
  Arms: Non Surgical Treatment
Procedure: Surgical — Initial surgical (stress incontinence surgery) treatment approach.
  Other Names: Surgical Treatment
  Arms: Surgical Treatment

SUMMARY:
The purpose of this study is to compare treatment outcomes for patients with mixed urinary incontinence (MUI) for whom therapy is initiated with surgery to those for whom therapy is initiated with non-surgical treatment. Women who are bothered by symptoms of both stress and urge incontinence will be randomly assigned to initiate treatment with a surgical (surgery for stress incontinence) vs. a non-surgical (drug and behavioral therapy) approach. Follow-up will be a minimum of 12 Months.

DETAILED DESCRIPTION:
The purpose of this study is to compare treatment outcomes for patients with mixed urinary incontinence (MUI) for whom therapy is initiated with surgery to those for whom therapy is initiated with non-surgical treatment. Women who are bothered by symptoms of both stress and urge incontinence will be randomly assigned to initiate treatment with a surgical (surgery for stress incontinence) vs. a non-surgical (drug and behavioral therapy) approach. Follow-up will be a minimum of 12 Months.

ELIGIBILITY:
Inclusion Criteria:

1. Female
2. Mixed UI as evidenced by stress and urge symptoms reported on MESA (either percent of urge-type symptoms ≥ the percent of stress-type symptoms or urge symptom score ≥7 if stress predominant) followed by report of "moderately" or "greatly"/"quite a bit" bothered to questions 2 and 3 of the 6-item Urinary Distress Index (UDI-6) or questions 16 and 17 of the 20-item Pelvic Fl;oor Distress Index (PFDI-20), respectively (See Appendix C)
3. Moderate or severe UI as evidenced by the corresponding response on the Patient Global Impression of Severity (PGI-S)
4. Incontinence symptoms present for at least (3) months*
5. Bladder capacity > 200cc (by any method)
6. Urodynamic Stress Incontinence
7. Eligible for both treatment interventions
8. Available to start intervention within 6 weeks
9. Negative urine dipstick (negative result = trace or less for leukocytes & nitrites)
10. Available for 12 months of follow-up and able to complete study assessments as per clinician judgment
11. Signed consent form

Exclusion Criteria:

1. Age <21 years*
2. Currently undergoing or recommended to undergo treatment of pelvic organ prolapse
3. Other indicated/planned concomitant surgery
4. Pregnant or has not completed child bearing*
5. <12 months post-partum*†
6. Active malignancy of cervix, uterus, fallopian tube(s) or ovary > Stage I, or bladder of any Stage
7. Current catheter use
8. Unevaluated hematuria
9. Participation in another trial that may influence the results of this study

   * Patient can be rescreened after respective time interval has been met. †"Partum" is defined as a delivery or other termination that occurs after 20 weeks gestation.

Min Age: 21 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 27 (Actual)
Dates: Start 2008-10; Primary Completion 2009-03 (Actual); Study Completion 2009-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ann Gormley, MD, Study Chair — Dartmouth-Hitchcock Medical Center
Locations (10):
- United States (10):
  - University of Alabama, Birmingham, Alabama
  - University of California, San Diego, California
  - Loyola University Medical Center, Maywood, Illinois
  - University of Maryland, Baltimore, Maryland
  - Oakwood Hospital/Cancer Center, Dearborn, Michigan
  - Beaumont Hospital, Royal Oak, Michigan
  - University of Pittsburgh, Pittsburgh, Pennsylvania
  - University of Texas Southwestern, Dallas, Texas
  - University of Texas Health Sciences Center, San Antonio, Texas
  - University of Utah, Salt Lake City, Utah

REFERENCES:
- [Background] Brubaker L, Moalli P, Richter HE, Albo M, Sirls L, Chai T, Kraus SR, Norton P, Chang D, Tennstedt SL. Challenges in designing a pragmatic clinical trial: the mixed incontinence -- medical or surgical approach (MIMOSA) trial experience. Clin Trials. 2009 Aug;6(4):355-64. doi: 10.1177/1740774509339239. Epub 2009 Jul 22. PMID 19625327
- See also: Urinary Incontinence Treatment Network (UITN) Public Website — http://www.uitn.net

RESULTS

PARTICIPANT FLOW:
Recruitment Details: 40 women were screened, 29 met eligibility criteria and 27 were enrolled between November, 2008 and March, 2009. The trial was terminated in March 2009 due to inadequate enrollment.
Pre-assignment Details: All enrolled participants were randomized.
Period: Overall Study
Arm/Group | Surgical Treatment | Non Surgical Treatment
Started | 13 | 14
Completed | 12 | 12
Not Completed | 1 | 2
Not completed — Lost to Follow-up | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Non Surgical Treatment: The non-surgical treatment will include two components:
  1. Pharmacological therapy with any FDA approved OAB drug in approved doses; and
  2. Behavioral therapy.
- Total: Total of all reporting groups
Arm/Group | Surgical Treatment | Non Surgical Treatment | Total
Number analyzed (Participants) | 13 | 14 | 27
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 11 | 19
  >=65 years | 5 | 3 | 8
Age Continuous [Mean (Standard Deviation); unit: years] | 53 (14) | 59 (14) | 56 (14)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 14 | 27
  Male | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 13 | 14 | 27

OUTCOME MEASURES:

1. Primary Outcome: Optimal Outcome of Treatment at 6 Months
Description: Composite measure defined as "much better" or "very much better" on Patient Global Impression of Improvement (PGI-I) and "normal" or "mild" on Patient Global Impression of Symptoms (PGI-S). PGI-I is a single item: "Circle the one answer that best describes your urinary tract condition now, compared to how it was before your incontinence treatment" with responses ranging from 1= "Very much better" to 7= "Very much worse." The PGI-S is a single item:; "Circle the one number that best describes how your urinary tract condition is now" with responses ranging from 1 = "Normal" to 4 "Severe".
Time Frame: 6 Months
Population: Participants who attended 6 month follow-up visit
Measure: Number; unit: participants
Arm/Group | Surgical Treatment | Non Surgical Treatment
Number analyzed (Participants) | 12 | 12
participants | 9 | 8
Statistical Analysis 1: Comparison: Surgical Treatment vs Non Surgical Treatment; Test type: Superiority or Other; p = 0.99, Fisher Exact; Difference of proportions = 0.08, 95% CI 2-sided [-0.28 to 0.44], Standard Error of Mean 0.19

2. Secondary Outcome: Optimal Outcome of Treatment at 3 Months
Description: Composite measure defined as "much better" or "very much better" om PGI-I and "normal" or "mild" on PGI-S. PGI-I is a single item: "Circle the one answer that best describes how your urinary tract condition is now, compared with how it was before your incontinence treatment" with responses ranging from 1="Very much better" to 7="Very much worse." PGI-S is a single items: "Circle the one number that best describes how your urinary tract condition is now" with responses ranging from 1="Normal" to 4="Severe."
Time Frame: 3 months
Population: Participants who attended 3 month follow-up visit
Measure: Number; unit: participants
Arm/Group | Surgical Treatment | Non Surgical Treatment
Number analyzed (Participants) | 10 | 12
participants | 7 | 3
Statistical Analysis 1: Comparison: Surgical Treatment vs Non Surgical Treatment; Test type: Superiority or Other; p = 0.08, Fisher Exact — Fisher's Exact Test of equality of percent meeting optimal outcome; difference of proportions = 0.45, 95% CI 2-sided [0.03 to 0.87], Standard Error of Mean 0.21

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Surgical Treatment | Non Surgical Treatment
Serious Adverse Events (participants affected / at risk) | 0/14 | 0/13
Other Adverse Events (participants affected / at risk) | 1/14 | 1/13
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Surgical Treatment (N=14) | Non Surgical Treatment (N=13)
Bladder perforation (Renal and urinary disorders) | 1 (1) | 0 (0)
Urinary retention (Renal and urinary disorders) | 0 (0) | 1 (1)

LIMITATIONS AND CAVEATS:
Early termination leading to small numbers of participants for data analysis.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other